CLINICAL TRIAL: NCT05183295
Title: Prospective Single Arm Medical Food Study to Evaluate a Standardized Nonessential Amino Acid Restriction (NEAAR) Medical Food for the Dietary Management of Metastatic Colorectal Cancer
Brief Title: Medical Food for the Dietary Management of Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn by Sponsor.
Sponsor: Faeth Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEAAR-002
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Nonessential Amino Acid Restriction (NEAAR) Medical Food (Experimental): All subjects will receive NEAAR medical food
  Interventions: Other: NEAAR Medical Food

INTERVENTIONS:
Other: NEAAR Medical Food — Standardized non-essential amino acid restricted medical food

SUMMARY:
This is a single arm study evaluating the tolerability and markers of colorectal cancer with a specially designed medical food restricted in specific amino acids for the dietary management of subjects with metastatic colorectal cancer. Subjects will be receiving two FDA approved second line drug therapies, fluoropyrimidine and oxaliplatin ± bevacizumab (FOLFIRI + BEV) that are routinely prescribed in combination for metastatic colorectal cancer as part of their routine care.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic and unresectable CRC.
2. Age ≥ 18 years.
3. ECOG Performance Status of ≤ 1.
4. Subject is not receiving any other cancer therapy. Subjects participating in surveys or observational studies are allowed.
5. Has failed treatment for fluoropyrimidine and oxaliplatin ± BEV.
6. FOLFIRI ± BEV therapy is prescribed for the subject per standard of care.
7. Subjects with measurable disease as determined by RECIST 1.1.
8. Must have acceptable organ function.

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (1500/μL).
   2. Platelet count ≥ 100 x 109/L.
   3. Hemoglobin ≥ 9 g/dL
   4. Activated partial thromboplastin time/international normalized ratio (aPTT/ INR) ≤ 1.5 x upper limit of normal (ULN) unless the subject is on anticoagulants in which case therapeutically acceptable values (as determined by the investigator) meet eligibility requirements.
   5. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤2.5 × ULN. In the case of known (i.e., radiological or biopsy documented) liver metastasis, serum transaminase levels must be ≤ 5 x ULN.
   6. Total serum bilirubin ≤ 1.5 x ULN (except for subjects with known Gilbert's Syndrome for which ≤ 3 x ULN is permitted).
   7. Serum creatinine < 2.0 x ULN and creatinine clearance ≥50 mL/min/1.73m2
   8. Serum albumin ≥3.5 mg/dL or ≥LLN, whichever is lower
9. Subjects must have available colorectal cancer (CRC) tissue samples from the most recently biopsied primary or metastatic site and provide consent for them to be obtained and analyzed.
10. Subjects must be willing to stop taking any supplements, herbal medicines, or alternative remedies or other prescribed or over the counter supplements for at least 1 week prior to Cycle 1 Day 1 of FOLFIRI ± BEV and through the NEAAR medical food period.

Exclusion Criteria:

1. Concomitant MSI-H/dMMR (Microsatellite Instability High/Deficient Mismatch Repair)
2. Anti-cancer chemotherapy or biologic therapy administered within 3 weeks prior to the first dose of fluoropyrimidine and irinotecan-based regimens . The exception is a single dose of radiation up to 8 Gray (equal to 800 RAD) with palliative intent for pain control up to 14 days before NEAAR medical food and return to baseline or ≤ Grade 1 toxicity associated with the radiation therapy.
3. More than one prior chemotherapy regimen administered in the metastatic setting.
4. Major surgery within 6 weeks prior to randomization.
5. Current brain metastasis.
6. Women who are pregnant or breastfeeding.
7. Gastrointestinal (GI) disorder(s) that, in the opinion of the investigator, would significantly impede the absorption of an oral agent (e.g., intestinal occlusion, active Crohn's disease, ulcerative colitis, extensive gastric, and small intestine resection). Exception: ostomy with normal daily stool output (<2L output).
8. Unable or unwilling to ingest the NEAAR medical food.
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure (CHF) Class II or higher according to the New York Heart Association (NYHA) Functional Classification, unstable angina pectoris, clinically significant cardiac arrhythmia, cardiac stent placement < 3 months prior to the NEAAR run in period, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements.

   1. Known active infection with Human Immunodeficiency Virus (HIV) and/or active infection with hepatitis B or C (patients who have had a hepatitis B virus [HBV] immunization are eligible).
   2. Clinically significant ascites or pleural effusions.
10. Diagnosis of another malignancy within the past 2 years (excluding a history of carcinoma in situ of the cervix, superficial non-melanoma skin cancer, superficial bladder cancer that has been adequately treated, or stage 1 prostate cancer that does not require treatment or requires only treatment with luteinizing hormone releasing hormone agonists or antagonists if initiated at least 30 days prior to beginning the NEAAR medical food).Any active disease condition that would render the protocol treatment dangerous or impair the ability of the patient to receive NEAAR
11. The following are exclusion criteria for patients who received SOC BEV:

    1. History of cardiac disease: congestive heart failure (CHF) Class II or higher according to the New York Heart Association (NYHA); active coronary artery disease, myocardial infarction within 6 months prior to study entry; unevaluated new onset angina within 3 months or unstable angina (angina symptoms at rest) or cardiac arrhythmias requiring antiarrhythmic therapy (beta blockers or digoxin are permitted).
    2. Current uncontrolled hypertension (systolic blood pressure [BP] > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management) or prior history of hypertensive crisis or hypertensive encephalopathy.
    3. History of arterial thrombotic or embolic events (within 6 months prior to study entry).
    4. Significant vascular disease (e.g., aortic aneurysm, aortic dissection, symptomatic peripheral vascular disease).
    5. Evidence of bleeding diathesis or clinically significant coagulopathy.
    6. Major surgical procedure (including open biopsy, significant traumatic injury, etc.) within 28 days, or anticipation of the need for major surgical procedure during the study, and minor surgical procedure (excluding placement of a vascular access device) within 7 days prior to study enrollment.
    7. Proteinuria at Screening as demonstrated by urinalysis with proteinuria ≥2+ (patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
    8. History of abdominal fistula, GI perforation, peptic ulcer, or intraabdominal abscess within 6 months.
    9. Ongoing serious, non-healing wound, ulcer, or bone fracture.
    10. Known hypersensitivity to any component of BEV.
    11. History of reversible posterior leukoencephalopathy syndrome (RPLS).
12. Comorbidity risk, that in the discretion of the investigator would make the subject a poor candidate for the NEAAR medical food.
13. A body mass index (BMI) <18.5 kg/m2 or >40 kg/m2, or serious or refractive cachexia or anorexia that, in the investigator's opinion, realistically prohibits subjects from having energy or appetite sufficient to reliably engage in a strict medical food regimen for an extended time.
14. Insulin-dependent or poorly controlled diabetes.
15. Subjects who must take medications that impact targeted amino acid levels
16. Inability or unwillingness to comply with study and/or follow-up procedures, or medical food modifications described in the protocol.
17. Untreated clinically significant hyperlipidemia per investigator.
18. Subjects with a condition (including gallbladder disease and/or fatty acid oxidation disorders or porphyria) where high-fat or fatty food is contraindicated.
19. Presence of any condition (e.g., persistent diarrhea) that renders the subject unable to satisfactorily chew, swallow, digest, absorb, or tolerate the majority of foods and liquids of the NEAAR medical food, especially high-fat foods such as oils, cream, and butter.
20. Taking or needs to take any protein or amino acid containing nutritional supplements (e.g., Ensure®).
21. Lack of physical integrity of the upper or lower gastrointestinal (GI) tract.
22. History of confirmed food allergy.
23. Unwillingness to consume small quantities of meat products and byproducts (for example fish sauce, bone marrow, chicken broth, etc.).
24. Diagnosis of previous or current eating disorder and/or disordered eating behaviors.
25. Diagnosed with Crohn's disease, ulcerative colitis, or gluten-sensitive enteropathy (Celiac disease).
26. Has previous epidermal growth factor receptor inhibitor (EGFRi) therapy or a combined fluoropyrimidine and irinotecan plus oxaliplatin-based regimen (e.g, FOLFIRINOX) in the first line treatment.
27. Is receiving or plans to receive a concomitant EGFRi inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Tolerability of the NEAAR medical food | Through study completion (average of 6 months)
  Rate of the most common Grade 3 and 4 adverse event (AE) related to the NEAAR medical food.

SECONDARY OUTCOMES:
Overall response rates | Through study completion (average of 6 months)
  Complete response and partial response per RECIST 1.1
Changes in biomarkers | Through study completion (average of 6 months)
  Absolute and relative change from baseline for disease biomarkers
Progression-free Survival | 6, 9 and 12 months
  Duration from radiographic documentation of disease to radiographic documentation of progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cerceck, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center